CLINICAL TRIAL: NCT02373059
Title: Examining the Use of a Shared Decision Making Tool With Pharmaceutical Care in Type 2 Diabetes
Brief Title: Shared Decision Making With Pharmaceutical Care
Acronym: SDMPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joseph R. Herges, Pharm.D., R.Ph., Doctor of Pharmacy, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-009665
Record Dates: First submitted 2015-02-16; First posted 2015-02-26 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmaceutical care with shared decision making (Experimental): Use of Diabetes Issue Cards Decision Aids
  Interventions: Other: Diabetes Issue Cards Decision Aids
- Usual Pharmaceutical care (Active Comparator): Usual Care
  Interventions: Other: Usual Pharmaceutical Care

INTERVENTIONS:
Other: Diabetes Issue Cards Decision Aids
  Arms: Pharmaceutical care with shared decision making
Other: Usual Pharmaceutical Care
  Arms: Usual Pharmaceutical care

SUMMARY:
A research study to enhance clinical discussion between patients and pharmacists using a shared decision making tool for type 2 diabetes or usual care.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Diagnosed with type II diabetes by ICD-9 code for more than one year
* HbA1c of 7%-9.5% within past 6 months
* Prescribed three or less anti-hyperglycemic medications as indicated by the medication list within the medical record

Exclusion Criteria:

* Prescribed insulin
* Pregnancy
* Appointment with provider within a month
* Appointment with provider within the last month
* Followed by endocrinology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Patient Involvement Questionnaire | Post-Visit up to 2 weeks

SECONDARY OUTCOMES:
Patient Knowledge regarding Diabetes treatments Questionnaire | post visit up to 2 weeks
Patient Medication Adherence Questionnaire | 1 month post visit

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic Kasson, Kasson, Minnesota, United States